CLINICAL TRIAL: NCT06851338
Title: Pediatric Down Syndrome Post-Approval Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Inspire Medical Systems, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-002
Record Dates: First submitted 2025-02-24; First posted 2025-02-28 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Pediatric Obstructive Sleep Apnea; Down Syndrome (DS)
Keywords: Pediatrics; OSA; Down Syndrome; Pediatrics OSA; Obstructive Sleep Apnea; Long-term follow-up; Post Approval Study; PAS
MeSH Terms: conditions — Down Syndrome; Sleep Apnea, Obstructive | interventions — Drug Delivery Systems

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Pediatric Postmarket Surveillance: Yes | US Export: Yes

ARMS (1):
- Pediatric subjects with Down syndrome undergoing Inspire UAS Implant (Experimental): This study is a prospective, multi-center, single-arm study of pediatric subjects (age 13-18) with Down syndrome who are undergoing implant of the Inspire Upper Airway Stimulation (UAS) system for the treatment of severe obstructive sleep apnea (OSA).
  Interventions: Device: Hypoglossal Nerve Stimulation

INTERVENTIONS:
Device: Hypoglossal Nerve Stimulation — Implant of Inspire Upper Airway Stimulation (UAS) system for treatment of obstructive sleep apnea (OSA) in the pediatric down syndrome population
  Other Names: Inspire Upper Airway Stimulation (UAS) System

SUMMARY:
The purpose of this Post Approval research study is to assess ongoing safety and effectiveness of the Inspire therapy in adolescents and young adults (age 13-18) with Down syndrome and severe sleep apnea. The objective of the study is to provide an ongoing safety and effectiveness assessment of the Inspire UAS System in the Pediatric Down syndrome population.

DETAILED DESCRIPTION:
This is a multi-center, prospective, single-arm study conducted under a common implant and follow-up protocol. The objective will be to follow sixty (60) adolescents (13 - 18), with Down Syndrome and severe sleep apnea for 5-years after undergoing implant of the Inspire Upper Airway Stimulation (UAS) system. The objective of the study is to provide an ongoing safety and effectiveness assessment of the Inspire UAS System in the Pediatrics Down Syndrome population.

Prior to implant subjects will be required to meet eligibility criteria that is based on an in-lab PSG, surgical consultation and drug induced sleep endoscopy, as well as other assessments. Subjects will also complete quality of life questionnaires.

During the 5-year follow-up period, data will be collected at the time of implant, and at multiple follow-up visits through five years post-implant. At each of these visits, safety information (adverse events), sleep data, therapy usage, and quality of life will be collected.

A total of sixty (60) subjects with even distribution across the age range will be implanted at a minimum of five (5) clinical centers in the US.

Subjects will conclude their participation in the study at the end of their 5 year follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has been diagnosed with Down syndrome;
2. Patient is 13-18 years of age;
3. Patient has been diagnosed with severe obstructive sleep apnea, with an AHI of ≥ 10 and ≤ 50 based on a recent (within 6 months of enrollment) qualified in-lab sleep study (PSG);
4. Patient has documented failure of, or intolerance to, positive airway pressure therapies (such as CPAP or BiPAP) despite attempts to improve compliance;
5. Patient is contraindicated for, or not effectively treated by, adenotonsillectomy;
6. Treatment of patient's OSA has followed standard of care in considering all other alternative/adjunctive therapies;
7. Patient, and their parents/guardians, is willing to have stimulation hardware permanently implanted, and be willing to participate in follow-up visits, postoperative in-lab sleep studies (PSGs), and questionnaire completion.

Exclusion Criteria:

1. Patient's recent PSG (within 6 months of enrollment) reports central + mixed apneas > 25% of the total apnea-hypopnea index (AHI);
2. Patient has any anatomical finding that would compromise the performance of upper airway stimulation, such as the presence of complete concentric collapse of the soft palate;
3. Patient has any condition or procedure that has compromised neurological control of the upper airway;
4. Patient, or their parent/guardian, is unable or does not have the necessary assistance to operate the patient remote;
5. Patient is pregnant or plans to become pregnant;
6. Patient has an implantable device that may be susceptible to unintended interaction with the Inspire system;
7. Patient will require magnetic resonance imaging (MRI) other than what is specified in the MR conditional labeling;
8. Patient has a terminal illness with life expectancy of less than 12 months;
9. Any other reason the investigator deems the patient is unfit for participation in the study.

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2030-05 (Estimated); Study Completion 2030-05 (Estimated)

PRIMARY OUTCOMES:
Safety Outcome Measure - Procedure and Device-related Adverse events | Implant through 5 Years
  Procedure-related and Device-related adverse events will be summarized by seriousness and severity. No formal hypothesis will be tested.
Effectiveness Outcome Measure - Comparison of Baseline and Annual Apnea-Hypopnea Index (AHI) | Baseline and Annually through 5 Years post-implant
  The AHI will be collected at each sleep study. This effectiveness measure will be reported as a comparison of baseline and annual (1-5 year) AHI.
  Descriptive statistics will be used to analyze this data. No formal hypothesis will be tested.

SECONDARY OUTCOMES:
Effectiveness Outcome Measure - Comparison of Baseline, 6 month, and Annual Epworth Sleepiness Scale for Children and Adolescents (ESS-CHAD) | Baseline, 6 months, and annually through 5-year post-implant
  The ESS-CHAD will be completed at baseline, as well as 6 months and annually (1-5 years) post-implant. The ESS-CHAD score at baseline compared to the ESS-CHAD score at each annual study visit will be reported.
  Descriptive statistics will be used to analyze this data. No formal hypothesis will be tested.
Effectiveness Outcome Measure - Comparison of Baseline and Annual Percent Time Oxygen Saturation < 90% (T90) | Baseline and Annually through 5-year post-implant
  Descriptive statistics will be used to analyze this data. No formal hypothesis will be tested.
Effectiveness Outcome Measure - Comparison of Baseline and Annual Oxygen Desaturation Index (ODI) | Baseline and Annually through 5 years post-implant
  The ODI will be collected during each sleep study. This effectiveness measure will be reported as a comparison of baseline and annual (1-5 year) ODI.
  Descriptive statistics will be used to analyze this data. No formal hypothesis will be tested.

OTHER OUTCOMES:
Ancillary Outcome Measure - Therapy Usage | 6 Months and Annually through 5 years post-implant
  Therapy usage, reported as hours per week and averaged into hours per night, will be used to quantify device use and adherence over time (6M, annually 1-5 years).
  Descriptive statistics will be used to analyze this data. No formal hypothesis will be tested.

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Children's Hospital Orange County, Orange, California
  - University of South Florida Morsani College of Medicine, Tampa, Florida
  - Northwell Cohen Children's Hospital, Queens, New York
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Baylor College of Medicine/ Texas Children's Hospital, Houston, Texas

IPD SHARING:
Plan to Share IPD: No